CLINICAL TRIAL: NCT04788511
Title: Effect of Semaglutide 2.4 mg Once Weekly on Function and Symptoms in Subjects With Obesity-related Heart Failure With Preserved Ejection Fraction
Brief Title: Research Study to Investigate How Well Semaglutide Works in People Living With Heart Failure and Obesity
Acronym: STEP-HFpEF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EX9536-4665; U1111-1243-4358 (Other: World Health Organization (WHO)); 2019-004452-11 (Registry Identifier: European Medicines Agency (EudraCT))
Record Dates: First submitted 2021-03-05; First posted 2021-03-09 (Actual); Results first posted 2024-06-11 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Semaglutide (Experimental): All participants will receive either semaglutide 2.4 mg once weekly or placebo once weekly as add-on to standard of care. During the first 16 weeks, the dose of semaglutide or placebo will be gradually escalated from 0.25 mg once weekly until target dose.
  Interventions: Drug: Semaglutide
- Placebo (semaglutide) (Placebo Comparator): All participants will receive either semaglutide 2.4 mg once weekly or placebo once weekly as add-on to standard of care. During the first 16 weeks, the dose of semaglutide or placebo will be gradually escalated from 0.25 mg once weekly until target dose.
  Interventions: Drug: Placebo (semaglutide)

INTERVENTIONS:
Drug: Semaglutide — Semaglutide will be injected into a skin fold, in the stomach, thigh or upper arm once a week at the same day of the week (to the extent possible) throughout the trial.
  Dose gradually escalated from 0.25 mg until target dose. The study will last for approximately 59 weeks.
  Arms: Semaglutide
Drug: Placebo (semaglutide) — Placebo will be injected into a skin fold, in the stomach, thigh or upper arm once a week at the same day of the week (to the extent possible) throughout the trial.
  The study will last for approximately 59 weeks.
  Arms: Placebo (semaglutide)

SUMMARY:
This study will look at how the participants daily life is affected by their heart failure. The study will also look at the change in participants body weight from the start to the end of the study. This is to compare the effect on heart failure symptoms and on body weight in people taking semaglutide (a new medicine) to people taking "dummy" medicine.

Participants will either get semaglutide or "dummy" medicine - which treatment participants get is decided by chance. Participants will need to take 1 injection once a week. The study medicine is injected with a thin needle in a skin fold in the stomach area, thigh or upper arm.

During the study participants will have talks with the study staff about healthy lifestyle choices including healthy food and physical activity.

The study will last for approximately 59 weeks. Participants will have 11 clinic visits and 1 phone call with the study doctor. Women: Women cannot take part if they are pregnant, breast-feeding or plan to become pregnant during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age above or equal to 18 years at the time of signing informed consent.
* Body mass index (BMI) greater than or equal to 30.0 kg/m^2
* New York Heart Association (NYHA) Class II-IV
* Left ventricular ejection fraction (LVEF) greater than or equal to 45 percentage at screening

Exclusion Criteria:

* A self-reported change in body weight greater than 5 kg (11 lbs) within 90 days before screening irrespective of medical records
* Haemoglobin A1c (HbA1c) greater than or equal to 6.5 percentage (48 mmol/mol) based on latest available value from medical records, no older than 3 months or if unavailable a local measurement at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 529 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2023-04-18 (Actual); Study Completion 2023-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 1452), Study Director — Novo Nordisk A/S
Locations (145):
- United States (50):
  - Eastern Shore Rsrch Inst, LLC, Fairhope, Alabama
  - National Heart Institute Cal, Beverly Hills, California
  - Keck Medical Center of USC - Outpatient Clinic, Los Angeles, California
  - Lundquist Inst-Biomed Innovtn, Torrance, California
  - Jacksonville Ctr For Clin Res, Jacksonville, Florida
  - First Coast Cardiovascular Institute, Jacksonville, Florida
  - Baptist Heart Specialists_Jacksonville, Jacksonville, Florida
  - CV Res Ctr of S Florida, Miami, Florida
  - Endeavor Health Clinical Operations-NCH, Arlington Heights, Illinois
  - University of Chicago Medicine, Chicago, Illinois
  - Endeavor Health Glenbook Hosp, Evanston, Illinois
  - Northwestern University_Chicago_0, Evanston, Illinois
  - Chicago Medical Research LLC, Hazel Crest, Illinois
  - Ascension St. Vincent Medical Group, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center_Kansas City, Kansas City, Kansas
  - Cotton-O'Neil Heart Center, Topeka, Kansas
  - The Research Group of Lexington LLC, Lexington, Kentucky
  - Baptist Health Louisville, Louisville, Kentucky
  - Baptist Health Madisonville, Inc, Madisonville, Kentucky
  - Grace Research, LLC, Bossier City, Louisiana
  - Heart Clinic of Hammond, Hammond, Louisiana
  - Grace Research, LLC_Shreveport, Shreveport, Louisiana
  - Louisiana Heart Center_Slidell, Slidell, Louisiana
  - Louisiana Heart Center, Slidell, Louisiana
  - Ascension Saint Agnes Heart Ca, Baltimore, Maryland
  - John Hopkins Hospital, Baltimore, Maryland
  - Henry Ford Hospital, Detroit, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Univ of Mississippi Med Ctr, Jackson, Mississippi
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - St Louis Heart & Vascular, P.C., St Louis, Missouri
  - Bryan Heart, Lincoln, Nebraska
  - CHI Health Clinic Cardiology (CUMC - Bergan Mercy), Omaha, Nebraska
  - St Francis Hospital Lindner Research Center, Greenvale, New York
  - NY Presbyt Hosp-W Cornell Med, New York, New York
  - Rochester General Hospital, Rochester, New York
  - Wake Forest School of Medicine, Winston-Salem, North Carolina
  - Lindner Center,Christ Hospital, Cincinnati, Ohio
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Hospital of University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical Univ of South Carolina_Charleston_0, Charleston, South Carolina
  - Sanford Health_Sioux Falls, Sioux Falls, South Dakota
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Utah School of Medicine, Salt Lake City, Utah
  - Cardiology Consultants of Danville Inc., Danville, Virginia
  - Virginia Heart, Falls Church, Virginia
  - Sentara Health Research Center, Norfolk, Virginia
  - Virginia Commonwealth University Health System, Richmond, Virginia
- Argentina (9):
  - CEMEDIC, CABA, Buenos Aires
  - Master Centre for Argentina, San Carlos de Bolívar, Buenos Aires
  - Centro de Investigación y Prevención Cardiovascular, CABA
  - CEMEDIC, CABA
  - Cardiología Palermo Duplicate, Ciudad Autónoma de Buenos Aire
  - Cardiología Palermo, Ciudad Autónoma de Buenos Aire
  - Instituto de Cardiología de Corrientes, Corrientes
  - Consultorio Integral de Atención al Diabético, Morón
  - Sanatorio Britanico S.A., Rosario, Santa Fe
- Australia (6):
  - The Canberra Hospital_Garran, Garran, Australian Capital Territory
  - Concord Repatriation General Hospital - Cardiology Department, Concord, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Royal Brisbane Hospital, Herston, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - Geelong Cardiology Research Unit, Geelong, Victoria
- Canada (14):
  - University of Calgary_Calgary, Calgary, Alberta
  - Univ of Alberta Hosp Edmonton, Edmonton, Alberta
  - North Shore Heart Centre, North Vancouver, British Columbia
  - SMH Cardiology Clinical Trials Inc., Surrey, British Columbia
  - St. Boniface Hospital, Winnipeg, Manitoba
  - Cambridge Cardiac Care Centre, Cambridge, Ontario
  - Partnrs Adv Cardio Eval (PACE), Newmarket, Ontario
  - North York Diagn & Cardiac Ctr, North York, Ontario
  - Oakville Cardiovascular Research LP, Oakville, Ontario
  - Dr James Cha, Oshawa, Ontario
  - Heart Health Institute Research, Inc., Scarborough Village, Ontario
  - Dr. Louis Yao, Weston, Ontario
  - Clinique Sante Cardio MC, Montreal, Quebec
  - Unv de Cardiologie et dePneum, Québec
- Czechia (9):
  - Nemocnice Jihlava Kardiologie, Jihlava
  - Nemocnice Jihlava, Jihlava
  - Vseobecna fakultni nemocnice a 1 LF UK v Praze, Prague
  - Všeobecná fakultní nemocnice v Praze, Prague
  - IKEM, Prague
  - MEDICON a.s., Prague
  - Poliklinika Holešovice VISIONARY - Medicon Pharm s.r.o., Prague
  - Nemocnice Slany Kardiologie, Slaný
  - Nemocnice Tábor a.s., Tábor
- Denmark (3):
  - Herlev og Gentofte Hospital, Hellerup, Capital Region
  - Aarhus Universitetshospital, Hjertesygdomme, Aarhus N
  - Kardiologisk Odense & Svendborg, Svendborg
- Germany (9):
  - Charité - Campus Virchow-Klinikum - Kardiologie, Angiologie und Intensivmedizin (CRU), Berlin
  - Cardiologicum Dresden und Pirna - MVZ "Am Felsenkeller" (Dresden), Dresden
  - Zentrum fuer klinische Studien Suedbrandenburg GmbH, Elsterwerda
  - MVZ CCB Frankfurt und Main-Taunus GbR, Frankfurt
  - Medical Center - University Of Freiburg, Freiburg im Breisgau
  - Universitätsklinikum Freiburg - Medical Center, Freiburg im Breisgau
  - Appel, Kassel
  - B. Braun Ambulantes Herzzentrum Kassel MVZ GmbH, Kassel
  - Universitatsklinikum Würzburg - Zentrum für Herzinsuffizienz, Würzburg
- Hungary (9):
  - Lausmed Kft., Baja, Bács-Kiskun county
  - Selye János Kórház, Komárom, Komárom-Esztergom
  - Szent Margit Rendelőintézet Nonprofit Kft., Budapest
  - Semmelweis Egyetem Szent Rókus Klinikai Tömb, Budapest
  - Gottsegen György Országos Kardiológiai Intézet, Budapest
  - Semmelweis Egyetem Városmajori Szív- és Érgyógyászat, Budapest
  - Jahn Ferenc Dél-pesti Kórház és Rendelőintézet, Budapest
  - Borsod-Abaúj-Zemplén Megyei Központi Kórház, Miskolc
  - Zala Megyei Szent Rafael Kórház, Zalaegerszeg
- Israel (5):
  - Hadassah Ein Karam MC - Cardio Department, Jerusalem
  - Western Galilee MC - Cardiology Department, Nahariya
  - Rabin MC Beilinson - Heart Failure Unit, Petah Tikva
  - Sourasky MC - Cardio Vascular Research Center, Tel Aviv
  - Sheba MC - Cardiology Clinical Research Unit, Tel Litwinsky
- Netherlands (6):
  - Gelre Ziekenhuizen Apeldoorn, Apeldoorn
  - Rode Kruis Ziekenhuis Beverwijk, Beverwijk
  - UMC Groningen, Groningen
  - Saxenburgh Medisch Centrum, Hardenberg
  - Frisius MC Leeuwarden, Leeuwarden
  - Bravis Ziekenhuis, Roosendaal
- Poland (6):
  - Malopolskie Centrum Sercowo-Naczyniowe, Chrzanów, Lesser Poland Voivodeship
  - Uniwersytecki Szpital Kliniczny w Bialymstoku K. Kardio, Bialystok, Podlaskie Voivodeship
  - Ind. Prak. Lek. w dziedz. Kardiologii lek. med. K. Cymerman, Gdynia, Pomeranian Voivodeship
  - Pro Familia Altera Sp. z o.o., Katowice, Silesian Voivodeship
  - I Katedra i Klinika Kardiologii WUM SPCSK, Warsaw
  - Uniwersytecki Szpital Kliniczny nr 2 Uniwersytetu Medycznego w Łodzi, Lodz, Łódź Voivodeship
- Spain (3):
  - Hospital Universitario La Zarzuela, Madrid
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela
  - Hospital Clinico Universitario de Valencia, Valencia
- United Kingdom (16):
  - Yeovil District Hospital - Clinical Research Unit, Yeovil, Somerset
  - St. Richards Hospital_Cardiology, Chichester, West Sussex
  - Barnet Hospital - Cardiology Department, Barnet
  - Southmead Hospital, Bristol
  - Ninewells Hospital, Dundee
  - Glasgow Clinical Research Facility, Glasgow
  - Glasgow Royal Infirmary, Glasgow
  - Queen Elizabeth University Hospital, Glasgow
  - Wycombe General Hospital, High Wycombe
  - Aintree University Hospital, Liverpool
  - University Hospital Aintree, Liverpool
  - Manchester Royal Infirmary, Manchester
  - Wythenshawe Hospital_North West Heart Centre, Manchester
  - Great Western Hospital, Swindon
  - Musgrove Park Hospital, Taunton
  - St George's Hospital, Tooting

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Background] Borlaug BA, Kitzman DW, Davies MJ, Rasmussen S, Barros E, Butler J, Einfeldt MN, Hovingh GK, Moller DV, Petrie MC, Shah SJ, Verma S, Abhayaratna W, Ahmed FZ, Chopra V, Ezekowitz J, Fu M, Ito H, Lelonek M, Melenovsky V, Nunez J, Perna E, Schou M, Senni M, van der Meer P, Von Lewinski D, Wolf D, Kosiborod MN. Semaglutide in HFpEF across obesity class and by body weight reduction: a prespecified analysis of the STEP-HFpEF trial. Nat Med. 2023 Sep;29(9):2358-2365. doi: 10.1038/s41591-023-02526-x. Epub 2023 Aug 27. PMID 37635157
- [Result] Kosiborod MN, Abildstrom SZ, Borlaug BA, Butler J, Rasmussen S, Davies M, Hovingh GK, Kitzman DW, Lindegaard ML, Moller DV, Shah SJ, Treppendahl MB, Verma S, Abhayaratna W, Ahmed FZ, Chopra V, Ezekowitz J, Fu M, Ito H, Lelonek M, Melenovsky V, Merkely B, Nunez J, Perna E, Schou M, Senni M, Sharma K, Van der Meer P, von Lewinski D, Wolf D, Petrie MC; STEP-HFpEF Trial Committees and Investigators. Semaglutide in Patients with Heart Failure with Preserved Ejection Fraction and Obesity. N Engl J Med. 2023 Sep 21;389(12):1069-1084. doi: 10.1056/NEJMoa2306963. Epub 2023 Aug 25. PMID 37622681
- [Derived] Kosiborod MN, Deanfield J, Pratley R, Borlaug BA, Butler J, Davies MJ, Emerson SS, Kahn SE, Kitzman DW, Lingvay I, Mahaffey KW, Petrie MC, Plutzky J, Rasmussen S, Ronnback C, Shah SJ, Verma S, Weeke PE, Lincoff AM; SELECT, FLOW, STEP-HFpEF, and STEP-HFpEF DM Trial Committees and Investigators. Semaglutide versus placebo in patients with heart failure and mildly reduced or preserved ejection fraction: a pooled analysis of the SELECT, FLOW, STEP-HFpEF, and STEP-HFpEF DM randomised trials. Lancet. 2024 Sep 7;404(10456):949-961. doi: 10.1016/S0140-6736(24)01643-X. Epub 2024 Aug 30. PMID 39222642
- [Derived] Shah SJ, Sharma K, Borlaug BA, Butler J, Davies M, Kitzman DW, Petrie MC, Verma S, Patel S, Chinnakondepalli KM, Einfeldt MN, Jensen TJ, Rasmussen S, Asleh R, Ben-Gal T, Kosiborod MN. Semaglutide and diuretic use in obesity-related heart failure with preserved ejection fraction: a pooled analysis of the STEP-HFpEF and STEP-HFpEF-DM trials. Eur Heart J. 2024 Sep 14;45(35):3254-3269. doi: 10.1093/eurheartj/ehae322. PMID 38739118
- [Derived] Butler J, Shah SJ, Petrie MC, Borlaug BA, Abildstrom SZ, Davies MJ, Hovingh GK, Kitzman DW, Moller DV, Verma S, Einfeldt MN, Lindegaard ML, Rasmussen S, Abhayaratna W, Ahmed FZ, Ben-Gal T, Chopra V, Ezekowitz JA, Fu M, Ito H, Lelonek M, Melenovsky V, Merkely B, Nunez J, Perna E, Schou M, Senni M, Sharma K, van der Meer P, Von Lewinski D, Wolf D, Kosiborod MN; STEP-HFpEF Trial Committees and Investigators. Semaglutide versus placebo in people with obesity-related heart failure with preserved ejection fraction: a pooled analysis of the STEP-HFpEF and STEP-HFpEF DM randomised trials. Lancet. 2024 Apr 27;403(10437):1635-1648. doi: 10.1016/S0140-6736(24)00469-0. Epub 2024 Apr 7. PMID 38599221
- [Derived] Butler J, Abildstrom SZ, Borlaug BA, Davies MJ, Kitzman DW, Petrie MC, Shah SJ, Verma S, Abhayaratna WP, Chopra V, Ezekowitz JA, Fu M, Ito H, Lelonek M, Nunez J, Perna E, Schou M, Senni M, van der Meer P, von Lewinski D, Wolf D, Altschul RL, Rasmussen S, Kosiborod MN. Semaglutide in Patients With Obesity and Heart Failure Across Mildly Reduced or Preserved Ejection Fraction. J Am Coll Cardiol. 2023 Nov 28;82(22):2087-2096. doi: 10.1016/j.jacc.2023.09.811. Epub 2023 Oct 8. PMID 37993201
- [Derived] Kosiborod MN, Verma S, Borlaug BA, Butler J, Davies MJ, Jon Jensen T, Rasmussen S, Erlang Marstrand P, Petrie MC, Shah SJ, Ito H, Schou M, Melenovsky V, Abhayaratna W, Kitzman DW; STEP-HFpEF Trial Committees and Investigators. Effects of Semaglutide on Symptoms, Function, and Quality of Life in Patients With Heart Failure With Preserved Ejection Fraction and Obesity: A Prespecified Analysis of the STEP-HFpEF Trial. Circulation. 2024 Jan 16;149(3):204-216. doi: 10.1161/CIRCULATIONAHA.123.067505. Epub 2023 Nov 12. PMID 37952180

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 83 sites in 13 countries, as follows: Argentina (6), Australia (5), Hungary (8), Czech Republic (5), Poland (6), Spain (3), Netherlands (6), Denmark (3), United States (16), Canada (4), Israel (5), Germany (7) and United Kingdom (9).
Groups:
- Semaglutide 2.4 mg: Participants with obesity (body mass index [BMI] greater than or equal to (≥) 30.0 kilogram per square meter (kg/m^2) related heart failure with preserved ejection fraction received semaglutide 2.4 milligrams (mg) once weekly by subcutaneous injection (in the abdomen, thigh or upper arm). Participants initially received 0.25 mg of semaglutide. The dose was then escalated every fourth week with increments of 0.25 mg for 16 weeks until the target dose of 2.4 mg was reached. The treatment period was 52 weeks.
- Placebo: Participants with obesity (BMI ≥30.0 kg/m^2) related heart failure with preserved ejection fraction received placebo once weekly by subcutaneous injection (in the abdomen, thigh or upper arm) for 52 weeks. The dose escalation and maintenance of placebo matched that of semaglutide.
Period: Overall Study
Arm/Group | Semaglutide 2.4 mg | Placebo
Started | 263 | 266
Full Analysis Set (FAS) | 263 | 266
Safety Analysis Set (SAS) | 263 | 266
Completed | 256 | 254
Not Completed | 7 | 12
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lost to Follow-up | 2 | 7
Not completed — Death | 3 | 4

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) population included all the randomized participants for this trial.
Groups:
- Semaglutide 2.4 mg: Participants with obesity (BMI ≥30.0 kg/m^2) related heart failure with preserved ejection fraction received semaglutide 2.4 mg once weekly by subcutaneous injection (in the abdomen, thigh or upper arm). Participants initially received 0.25 mg of semaglutide. The dose was then escalated every fourth week with increments of 0.25 mg for 16 weeks until the target dose of 2.4 mg was reached. The treatment period was 52 weeks.
- Total: Total of all reporting groups
Arm/Group | Semaglutide 2.4 mg | Placebo | Total
Number analyzed (Participants) | 263 | 266 | 529
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (9) | 68 (10) | 68 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 149 | 148 | 297
  Male | 114 | 118 | 232
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 21 | 36
  Not Hispanic or Latino | 248 | 245 | 493
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 13 | 21
  White | 255 | 252 | 507
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Kansas City Cardiomyopathy Questionnaire Clinical Summary Score (KCCQ-CSS)
Description: The KCCQ is a standardized 23-item, self-administered instrument that quantifies heart failure symptoms (frequency, severity, and recent change), physical limitation, quality of life, and social limitation. The overall summary score and all domains have been independently demonstrated to be valid, reliable, and responsive to clinical change. KCCQ-CSS includes the symptom and physical limitation domains of the KCCQ. Scores are transformed to a range of 0-100, in which higher scores reflect better health status. The outcome measure was evaluated based on the data from in-trial period. In-trial period was defined as the uninterrupted time interval from date of randomization to date of last contact with trial site.
Time Frame: From baseline (week 0) to end of treatment (week 52)
Population: FAS included all the randomized participants for this trial. Here, Overall Number of Participants Analyzed" signifies those participants who had an observed value at week 52.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 243 | 237
Score on a scale | 16.8 (17.9) | 10.3 (17.3)
Statistical Analysis 1: Comparison: Semaglutide 2.4 mg vs Placebo; The responses at week 52 were analyzed using an analysis of covariance model with randomized treatment and stratification (BMI<35.0 kg/m^2, BMI>=35.0 kg/m^2) as factors and baseline KCCQ-CSS as covariate. The analysis was based on the in-trial period using the FAS population. Missing observations at week 52 were multiple (x1000) imputed from retrieved participants of the same randomized treatment arm; Test type: Superiority; p < 0.0001, ANCOVA; Estimated Treatment Difference = 7.8, 95% CI 2-sided [4.8 to 10.9]

2. Primary Outcome: Change in Body Weight
Description: Change in body weight from baseline (week 0) to end of treatment (week 52) is presented. The outcome measure was evaluated based on the data from in-trial period. In-trial period was defined as the uninterrupted time interval from date of randomization to date of last contact with trial site.
Time Frame: From baseline (week 0) to end of treatment (week 52)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of body weight
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 246 | 242
Percentage of body weight | -13.9 (8.1) | -2.5 (5.6)
Statistical Analysis 1: Comparison: Semaglutide 2.4 mg vs Placebo; The responses were analyzed using an analysis of covariance model with randomized treatment and stratification (BMI<35.0 kg/m^2, BMI>=35.0 kg/m^2) as factors and baseline body weight (kg) as covariate. The analysis was based on the in-trial period using the FAS population. Missing observations at week 52 were multiple (x1000) imputed from retrieved participants of the same randomized treatment arm; Test type: Superiority; p < 0.0001, ANCOVA; Estimated Treatment Difference = -10.7, 95% CI 2-sided [-11.9 to -9.4]

3. Secondary Outcome: Change in Six-minute Walking Distance (6MWD)
Description: Observed mean change from baseline (week 0) in 6 minutes walking distance (6MWD) test to end of treatment (week 52) is presented. The 6MWD is a common test of functional exercise capacity that assesses the distance a participant can walk in 6 minutes. The outcome measure was evaluated based on the data from in-trial period. In-trial period was defined as the uninterrupted time interval from date of randomization to date of last contact with trial site.
Time Frame: From baseline (week 0) to end of treatment (week 52)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 240 | 225
Meters | 23.5 (59.2) | 5.8 (62.7)

4. Secondary Outcome: The Hierarchical Composite Endpoint: Percentage of Wins of Participant Pairs
Description: The hierarchical composite outcome measure from baseline (week 0) to end of study (week 57) consists of the components: time to all-cause death, number of heart failure events requiring hospitalization or urgent heart failure visit, time to first heart failure event requiring hospitalization or urgent heart failure visit, difference at least 15 in KCCQ CSS change from baseline to 52 weeks, difference at least 10 in KCCQ CSS change from baseline to 52 weeks, difference at least 5 in KCCQ CSS change from baseline to 52 weeks and difference at least 30 meters in six-minute walking distance change from baseline to 52 weeks. It was analyzed by the win-ratio approach using all participants pairs across treatment groups. Overall summary of wins in each treatment group is presented. The outcome measure was evaluated based on the data from in-trial period. In-trial period was defined as uninterrupted time interval from date of randomization to date of last contact with trial site.
Time Frame: From baseline (week 0) to end of study (week 57)
Population: FAS included all the randomized participants for this trial.
Measure: Number; unit: Percentages of wins of participant pairs
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 263 | 266
Percentages of wins of participant pairs | 60.1 | 34.9

5. Secondary Outcome: Change in C-Reactive Protein (CRP): Ratio to Baseline
Description: Change in high sensitivity C-reactive protein measured in ratio of C-reactive protein to baseline (week -2) at end of treatment (week 52) is presented. The outcome measure was evaluated based on the data from in-trial period. In-trial period was defined as the uninterrupted time interval from date of randomization to date of last contact with trial site.
Time Frame: From baseline (week -2) to end of treatment (week 52)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of C-reactive protein
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 241 | 243
Ratio of C-reactive protein | 0.55 (121.5) | 0.92 (105.3)

6. Secondary Outcome: Percentage of Participants Achieving 10 Percent (%) Weight Loss (Yes/No)
Description: Percentage of participants who achieved 10% weight loss (yes/no) from baseline (week 0) to end of treatment (week 52) is presented. In the reported data, 'Yes' infers percentage of participants who have achieved 10% weight loss whereas 'No' infers percentage of participants who have not achieved 10% weight loss. The outcome measure was evaluated based on the data from in-trial period. In-trial period was defined as the uninterrupted time interval from date of randomization to date of last contact with trial site.
Time Frame: From baseline (week 0) to end of treatment (week 52)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 246 | 242
Percentage of participants
  No | 34.1 | 90.5
  Yes | 65.9 | 9.5

7. Secondary Outcome: Percentage of Participants Achieving 15% Weight Loss (Yes/No)
Description: Percentage of participants who achieved 15% weight loss (yes/no) from baseline (week 0) to end of treatment (week 52) is presented. In the reported data, 'Yes' infers percentage of participants who have achieved 15% weight loss whereas 'No' infers percentage of participants who have not achieved 15% weight loss. The outcome measure was evaluated based on the data from in-trial period. In-trial period was defined as the uninterrupted time interval from date of randomization to date of last contact with trial site.
Time Frame: From baseline (week 0) to end of treatment (week 52)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 246 | 242
Percentage of participants
  No | 56.1 | 97.9
  Yes | 43.9 | 2.1

8. Secondary Outcome: Percentage of Participants Achieving 20% Weight Loss (Yes/No)
Description: Percentage of participants who achieved 20% weight loss (yes/no) from baseline (week 0) to end of treatment (week 52) is presented. In the reported data, 'Yes' infers percentage of participants who have achieved 20% weight loss whereas 'No' infers percentage of participants who have not achieved 20% weight loss The outcome measure was evaluated based on the data from in-trial period. In-trial period was defined as the uninterrupted time interval from date of randomization to date of last contact with trial site.
Time Frame: From baseline (week 0) to end of treatment (week 52)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 246 | 242
Percentage of participants
  No | 76.4 | 99.6
  Yes | 23.6 | 0.4

9. Secondary Outcome: Percentage of Participants Improving 5 Points or More in KCCQ Clinical Summary Score (Yes/No)
Description: Percentage of participants improving 5 points or more in KCCQ-CSS from baseline to end of treatment is presented. The KCCQ is standardized 23-item, self-administered instrument that quantifies heart failure symptoms(frequency, severity, and recent change), physical limitation, quality of life, and social limitation. KCCQ-CSS includes the symptom and physical limitation domains of the KCCQ. Scores are transformed to range of 0-100, in which higher scores reflect better health status. In the reported data, 'Yes' infers percentage of participants who have improved 5 points or more in score whereas 'No' infers percentage of participants who have not improved 5 points or more in score. The outcome measure was evaluated based on the data from in-trial period. In-trial period was defined as the uninterrupted time interval from date of randomization to date of last contact with trial site.
Time Frame: From baseline (week 0) to end of treatment (week 52)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 243 | 237
Percentage of participants
  No | 24.7 | 36.3
  Yes | 75.3 | 63.7

10. Secondary Outcome: Percentage of Participants Improving 10 Points or More in KCCQ Clinical Summary Score (Yes/No)
Description: Percentage of participants improving 10 points or more in KCCQ-CSS from baseline to end of treatment is presented. The KCCQ is standardized 23-item, self-administered instrument that quantifies heart failure symptoms(frequency, severity, and recent change), physical limitation, quality of life, and social limitation. KCCQ-CSS includes the symptom and physical limitation domains of the KCCQ. Scores are transformed to range of 0-100, in which higher scores reflect better health status. In reported data, 'Yes' infers percentage of participants who have improved 5 points or more in score whereas 'No' infers percentage of participants who have not improved 10 points or more in score. The outcome measure was evaluated based on the data from in-trial period. In-trial period was defined as the uninterrupted time interval from date of randomization to date of last contact with trial site.
Time Frame: From baseline (week 0) to end of treatment (week 52)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 243 | 237
Percentage of participants
  No | 36.6 | 51.5
  Yes | 63.4 | 48.5

11. Secondary Outcome: Change in KCCQ Overall Summary Score (KCCQ-OSS)
Description: The KCCQ is a standardized 23-item, self-administered instrument that quantifies heart failure symptoms (frequency, severity, and recent change), physical limitation, quality of life, and social limitation. The overall summary score and all domains have been independently demonstrated to be valid, reliable, and responsive to clinical change. KCCQ-CSS includes the symptom and physical limitation domains of the KCCQ while KCCQ-OSS includes the symptom, physical limitation, quality of life, and social limitation domains. Scores are transformed to a range of 0-100, in which higher scores reflect better health status. The outcome measure was evaluated based on the data from in-trial period. In-trial period was defined as the uninterrupted time interval from date of randomization to date of last contact with trial site.
Time Frame: From baseline (week 0) to end of treatment (week 52)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 243 | 237
Score on a scale | 16.8 (18.3) | 10.9 (17.5)

12. Secondary Outcome: Percentage of Participants Achieving Threshold for Clinically Meaningful Within-participants Change in KCCQ-CSS (PGI-S)
Description: The patient global impression of status (PGI-S) for KCCQ was used to rate participants' symptoms of heart failure using 4-category ordinal scale (no symptoms, mild, moderate, severe). KCCQ is standardized 23-item, self-administered instrument that quantifies heart failure symptoms (frequency, severity, and recent change), physical limitation, quality of life, and social limitation. OSS and all domains have been independently demonstrated to be valid, reliable, and responsive to clinical change. KCCQ-CSS includes symptom and physical limitation domains of the KCCQ. Scores are transformed to range of 0-100, in which higher scores reflect better health status. Outcome measure was evaluated based on data from in-trial period. In-trial period was defined as uninterrupted time interval from date of randomization to date of last contact with trial site. The threshold was defined as mean change in KCCQ-CSS in those participants with one-category improvement in PGI-S from baseline to week 52.
Time Frame: From baseline (week 0) to end of treatment (week 52)
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 243 | 237
Percentage of Participants | 43.2 | 32.5

13. Secondary Outcome: Percentage of Participants Achieving Threshold for Clinically Meaningful Within-participants Change in 6MWD (PGI-S)
Description: Observed mean change from baseline in 6 minutes walking distance (6MWD) test using PGI-S is evaluated for this outcome measure. The 6MWD is a common test of functional exercise capacity that assesses the distance a participant can walk in 6 minutes. The outcome measure was evaluated based on the data from in-trial period. In-trial period was defined as the uninterrupted time interval from date of randomization to date of last contact with trial site. The threshold was defined as the mean change in 6MWD in those participants with an one-category improvement in PGI-S from baseline to week 52.
Time Frame: From baseline (week 0) to end of treatment (week 52)
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 240 | 225
Percentage of Participants | 42.5 | 28.0

14. Secondary Outcome: Change in Systolic Blood Pressure (SBP)
Description: Observed mean change in systolic blood pressure from baseline (week -2) to end of treatment (week 52) is presented. The outcome measure was evaluated based on the data from in-trial period. In-trial period was defined as the uninterrupted time interval from date of randomization to date of last contact with trial site.
Time Frame: From baseline (week -2) to end of treatment (week 52)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimetre of mercury (mmHg)
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 246 | 243
millimetre of mercury (mmHg) | -6.4 (19.0) | -1.1 (17.5)

15. Secondary Outcome: Change in Waist Circumference
Description: Change waist circumference from baseline (week 0) to end of the treatment (visit 52) presented. Waist circumference is defined as the abdominal circumference located midway between the lower rib margin and the iliac crest. Measurement must be obtained in standing position with a non-stretchable measuring tape and to the nearest cm or inch. The tape should touch the skin but not compress soft tissue and twists in the tape should be avoided. The participant should be asked to breathe normally. The same measuring tape should be used throughout the trial. The outcome measure was evaluated based on the data from in-trial period. In-trial period was defined as the uninterrupted time interval from date of randomization to date of last contact with trial site.
Time Frame: From baseline (week 0) to end of treatment (visit 52)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Centimeter
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 246 | 240
Centimeter | -12.0 (8.5) | -2.8 (7.4)

ADVERSE EVENTS:
Time Frame: From baseline (week 0) to end of trial (week 57)
Description: All presented adverse events are treatment-emergent adverse events (TEAEs). A TEAEs was defined as an event that had onset during the on-treatment period (date of first trial product administration to date of last trial product administration excluding potential off-treatment time intervals triggered by at least five consecutive missed doses). SAS included all the participants who randomly assigned to trial treatment and who took at least one dose of trial product.
Arm/Group | Semaglutide 2.4 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 3/263 | 4/266
Serious Adverse Events (participants affected / at risk) | 35/263 | 71/266
Other Adverse Events (participants affected / at risk) | 93/263 | 57/266
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide 2.4 mg (N=263) | Placebo (N=266)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal wall haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 5 (6) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Amyloidosis (Immune system disorders) | 1 (1) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 2 (2) | 0 (0)
Arterial injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 9 (12)
Atrial flutter (Cardiac disorders) | 0 (0) | 3 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 3 (3)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 12 (13)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 3 (3)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 3 (4)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 2 (2)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 2 (2)
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 1 (1)
Embolic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Endometritis (Infections and infestations) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 1 (3)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Haematoma evacuation (Surgical and medical procedures) | 0 (0) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hydrocele (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemic unconsciousness (Nervous system disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 2 (2) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 2 (2)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 1 (1)
Medical observation (Investigations) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 2 (2)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Obstructive pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinovirus infection (Infections and infestations) | 0 (0) | 1 (1)
SARS-CoV-2 test positive (Investigations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Spondylitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Superficial spreading melanoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 1 (1)
Tricuspid valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Uterine polyp (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 2 (3)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide 2.4 mg (N=263) | Placebo (N=266)
COVID-19 (Infections and infestations) | 36 (36) | 41 (43)
Constipation (Gastrointestinal disorders) | 17 (18) | 7 (8)
Diarrhoea (Gastrointestinal disorders) | 24 (28) | 10 (16)
Nausea (Gastrointestinal disorders) | 45 (51) | 7 (8)
Vomiting (Gastrointestinal disorders) | 17 (22) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2023-06-21): https://cdn.clinicaltrials.gov/large-docs/11/NCT04788511/Prot_002.pdf
  • Statistical Analysis Plan (2022-12-01): https://cdn.clinicaltrials.gov/large-docs/11/NCT04788511/SAP_003.pdf